CLINICAL TRIAL: NCT05218564
Title: Air as a Placebo: Increasing the Respiratory Performance of People With COPD Through Simple Expectations of Improvement. An Experimental, Randomised, Two-arm, Counterbalanced Study With Three Data Collection Sessions.
Brief Title: Air as a Placebo: Increasing the Respiratory Performance of People With COPD Through Simple Expectations of Improvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Paolo Banfi, Head of U.O.C. Cardio-Respiratory Rehabilitation, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FDG_Placebo_COPD
Record Dates: First submitted 2021-12-28; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Placebo; Oxygen therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: It is foreseen that the professional (Psychologist other than the one involved in the administration of the tests inherent to the assessment), once the patient has been identified, proposed the study and the readiness to manage the eventual episode of acute respiratory infection, and obtained his consent, will use the results of the above-mentioned system to assign the participant to one of the two groups and therefore to the order of conditions. In this way, the physiotherapist performing the planned treatment, the psychologist involved in administering the psychological assessment and the physician performing the respiratory function tests will be excluded from the randomisation process and blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1, consisting of participants with COPD and usually using O2 (Experimental): In this group, in addition to the standard care, the participant undergoes the 6 Minute Walking Test (6MWT) using compressed medical air (RA) cylinders, believing that there is oxygen (O2) inside the cylinder. The same, then, in addition to the standard care, is subjected to the execution of the 6 Minute Walking Test (6MWT), thanks to the use of cylinders of Oxygen (O2), believing that inside the cylinder there is Oxygen (O2). The sequence of this group will then be characterised as follows: ABC (A=Baseline, B=Air, C=Oxygen).
  Interventions: Other: Compressed Medical Air
- Group 2, consisting of participants with COPD and usually not using O2 (Placebo Comparator): In this group, in addition to standard care, the participant is given the 6 Minute Walking Test (6MWT) using oxygen (O2) cylinders, believing that there is oxygen (O2) inside the cylinder. Next, the participant undergoes the 6 Minute Walking Test (6MWT), using compressed medical air (RA) cylinders, believing that there is oxygen (O2) inside the cylinder. The sequence of this group will be characterised as follows: ACB (A=Baseline, B=Air, C=Oxygen).
  Interventions: Drug: Oxygen Therapy

INTERVENTIONS:
Drug: Oxygen Therapy — During the 6 Minute Walking Test (6MWT), the participant will be required to walk as fast as possible on a flat, straight surface on the ward (e.g. corridor) in six minutes, including as many breaks as he/she deems necessary. The performance of this test will be monitored continuously by a Respiratory Physiotherapist and will include the presence of a Physician, who will be ready to assist as needed. The sequence of use of compressed medical air and oxygen used during the 6MWT in the first group will then be characterised as follows: ABC (A=Baseline, B=Air, C=Oxygen). The sequence of the second group will be characterised as follows: ACB (A=Baseline, B=Air, C=Oxygen).
  Arms: Group 2, consisting of participants with COPD and usually not using O2
Other: Compressed Medical Air — During the 6 Minute Walking Test (6MWT), the participant will be required to walk as fast as possible on a flat, straight surface on the ward (e.g. corridor) in six minutes, including as many breaks as he/she deems necessary. The performance of this test will be monitored continuously by a Respiratory Physiotherapist and will include the presence of a Physician, who will be ready to assist as needed. The sequence of use of compressed medical air and oxygen used during the 6MWT in the first group will then be characterised as follows: ABC (A=Baseline, B=Air, C=Oxygen). The sequence of the second group will be characterised as follows: ACB (A=Baseline, B=Air, C=Oxygen).
  Other Names: Placebo
  Arms: Group 1, consisting of participants with COPD and usually using O2

SUMMARY:
COPD (Chronic Obstructive Pulmonary Disease) is a disease of the respiratory system characterised by irreversible airway obstruction of varying severity. The disease (known as COPD, Chronic Obstructive Pulmonary Disease) is progressive and is associated with a state of chronic inflammation of the lung tissue, which leads to a real remodelling of the bronchi causing a significant reduction in airway flow. Among the possible treatments, while the placebo is considered as an inert treatment, lacking any intrinsic therapeutic properties, there is evidence in the literature that not all placebos are equivalent and some are more effective than others, as for example in the case of migraine or osteoarthritis. The differences found between different types of placebos (e.g. oral, subcutaneous, intra-articular...) indicate that placebos are not inert but rather consist of multiple psychosocial elements that are part of the ritual of the therapeutic act. This is also the context for the studies by Lacasse et al. (for the International Nocturnal Oxygen (INOX) Research Group et al., 2017) and Jarosh et al., who investigated the effects of oxygen therapy both during sleep and during the course of daily life, studying its influences through the use of placebo in patients suffering from hypoxemia. However, in the literature, there are no studies investigating the role of oxygen (O2) during the performance of a test such as the Walking Test, otherwise known as the 6 Minute Walking Test (6MWT) compared with a placebo in patients with Chronic Obstructive Pulmonary Disease (COPD), nor whether the use of the latter would lead to comparable results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily agree to participate in the study;
* Subjects with moderate-grade Chronic Obstructive Pulmonary Disease (COPD) (GOLD 2-50% ≤ FEV1 <80% of predicted) according to GOLD criteria;
* Subjects undergoing treatment with oxygen therapy and non-smokers;
* Ex-smokers
* Outpatients and inpatients

Exclusion Criteria:

* Refusal of Informed Consent
* Severe cognitive impairment, detected by administration of the Mini Mental Status Examination Test (MMSE)
* Pregnancy
* Patients with oncological or psychiatric pathologies
* Main immunodepression

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Metres covered during 6 Minute Walking Test (6MWT) | Changes from baseline at the metres covered after the completion of the 6MWT performed using oxygen or compressed medical air. Up to 1 hour and half
  Distance in metres during the 6 Minute Walking Test (6MWT)

SECONDARY OUTCOMES:
Feeling of fatigue, as measured by the Fatigue Severity Scale (FSS) | Changes from baseline at the FSS after the completion of the 6MWT performed using oxygen or compressed medical air. Up to 1 hour and half
  Feeling of fatigue, as measured by the Fatigue Severity Scale (FSS). The items are scored on a 7 point scale with 1=strongly disagree and 7=strongly agree. The minimum score=9 and maximum score possible=63. Higher the score=greater fatigue severity.
VAS Dyspnoea, measured by the British Medical Research Council's Modified Questionnaire (mMRC) | Change from baseline at the dyspnoea after the completion of the 6MWT performed using oxygen or compressed medical air. Up to 1 hour and half
  VAS Dyspnoea, measured by the British Medical Research Council's Modified Questionnaire (mMRC). The mMRC breathlessness scale ranges from grade 0 to 4.
Saturation (SpO2) | Change from baseline at 3':30'' and at 6':00'' of the 6 Minute Walking Test (6MWT)
  Saturation (SpO2)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Santa Maria Nascente, Fondazione Don Carlo Gnocchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bannuru RR, McAlindon TE, Sullivan MC, Wong JB, Kent DM, Schmid CH. Effectiveness and Implications of Alternative Placebo Treatments: A Systematic Review and Network Meta-analysis of Osteoarthritis Trials. Ann Intern Med. 2015 Sep 1;163(5):365-72. doi: 10.7326/M15-0623. PMID 26215539
- [Result] Barnes PJ. Chronic obstructive pulmonary disease: a growing but neglected global epidemic. PLoS Med. 2007 May;4(5):e112. doi: 10.1371/journal.pmed.0040112. PMID 17503959
- [Result] Benedetti F. Placebo and the new physiology of the doctor-patient relationship. Physiol Rev. 2013 Jul;93(3):1207-46. doi: 10.1152/physrev.00043.2012. PMID 23899563
- [Result] Benedetti F. Placebo effects: from the neurobiological paradigm to translational implications. Neuron. 2014 Nov 5;84(3):623-37. doi: 10.1016/j.neuron.2014.10.023. Epub 2014 Nov 5. PMID 25442940
- [Result] Benedetti F, Dogue S. Different Placebos, Different Mechanisms, Different Outcomes: Lessons for Clinical Trials. PLoS One. 2015 Nov 4;10(11):e0140967. doi: 10.1371/journal.pone.0140967. eCollection 2015. PMID 26536471
- [Result] Benedetti F, Durando J, Giudetti L, Pampallona A, Vighetti S. High-altitude headache: the effects of real vs sham oxygen administration. Pain. 2015 Nov;156(11):2326-2336. doi: 10.1097/j.pain.0000000000000288. PMID 26164587
- [Result] Benedetti F, Durando J, Vighetti S. Nocebo and placebo modulation of hypobaric hypoxia headache involves the cyclooxygenase-prostaglandins pathway. Pain. 2014 May;155(5):921-928. doi: 10.1016/j.pain.2014.01.016. Epub 2014 Jan 21. PMID 24462931
- [Result] Berry MJ, Rejeski WJ, Adair NE, Zaccaro D. Exercise rehabilitation and chronic obstructive pulmonary disease stage. Am J Respir Crit Care Med. 1999 Oct;160(4):1248-53. doi: 10.1164/ajrccm.160.4.9901014. PMID 10508815
- [Result] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Result] Blinderman CD, Homel P, Billings JA, Tennstedt S, Portenoy RK. Symptom distress and quality of life in patients with advanced chronic obstructive pulmonary disease. J Pain Symptom Manage. 2009 Jul;38(1):115-23. doi: 10.1016/j.jpainsymman.2008.07.006. Epub 2009 Feb 20. PMID 19232893
- [Result] de Craen AJ, Tijssen JG, de Gans J, Kleijnen J. Placebo effect in the acute treatment of migraine: subcutaneous placebos are better than oral placebos. J Neurol. 2000 Mar;247(3):183-8. doi: 10.1007/s004150050560. PMID 10787112
- [Result] Dowson CA, Kuijer RG, Mulder RT. Anxiety and self-management behaviour in chronic obstructive pulmonary disease: what has been learned? Chron Respir Dis. 2004;1(4):213-20. doi: 10.1191/1479972304cd032rs. PMID 16281648
- [Result] Lacasse Y, Bernard S, Series F, Nguyen VH, Bourbeau J, Aaron S, Maltais F; International Nocturnal Oxygen (INOX) Research Group. Multi-center, randomized, placebo-controlled trial of nocturnal oxygen therapy in chronic obstructive pulmonary disease: a study protocol for the INOX trial. BMC Pulm Med. 2017 Jan 9;17(1):8. doi: 10.1186/s12890-016-0343-9. PMID 28069009
- [Result] Jarosch I, Gloeckl R, Damm E, Schwedhelm AL, Buhrow D, Jerrentrup A, Spruit MA, Kenn K. Short-term Effects of Supplemental Oxygen on 6-Min Walk Test Outcomes in Patients With COPD: A Randomized, Placebo-Controlled, Single-blind, Crossover Trial. Chest. 2017 Apr;151(4):795-803. doi: 10.1016/j.chest.2016.11.044. Epub 2016 Dec 8. PMID 27940278
- [Result] Kong J, Spaeth R, Cook A, Kirsch I, Claggett B, Vangel M, Gollub RL, Smoller JW, Kaptchuk TJ. Are all placebo effects equal? Placebo pills, sham acupuncture, cue conditioning and their association. PLoS One. 2013 Jul 31;8(7):e67485. doi: 10.1371/journal.pone.0067485. Print 2013. PMID 23935833
- [Result] Wong CJ, Goodridge D, Marciniuk DD, Rennie D. Fatigue in patients with COPD participating in a pulmonary rehabilitation program. Int J Chron Obstruct Pulmon Dis. 2010 Oct 5;5:319-26. doi: 10.2147/COPD.S12321. PMID 21037955